CLINICAL TRIAL: NCT05694819
Title: Phase II Study of Darolutamide (ODM-201) in Patients With Androgen Receptor-positive Salivary Gland Carcinoma (Discovary Study)
Brief Title: Darolutamide in Patients With Androgen Receptor-Positive Salivary Gland Carcinoma (DISCOVARY)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center Hospital East (Other)
Collaborators: Bayer Yakuhin, Ltd. (Industry)
Responsible Party: Principal Investigator, Makoto Tahara, Chief, Department of Head and Neck Medical Oncology, National Cancer Center Hospital East
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: YCU19003; jRCT2031190241 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Salivary Gland Cancer
Keywords: Androgen receptor (AR)-positive; Salivary gland carcinoma; Darolutamide; luteinizing hormone-releasing hormone (LH-RH) analogue
MeSH Terms: conditions — Salivary Gland Neoplasms; Bulbo-Spinal Atrophy, X-Linked | interventions — darolutamide; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Darolutamide monotherapy (Experimental): Targeted patients: 24
  Interventions: Drug: Darolutamide
- Darolutamide plus Goserelin (Experimental): Targeted patients: 32
  Interventions: Drug: Darolutamide; Drug: Goserelin

INTERVENTIONS:
Drug: Darolutamide — Darolutamide at a dose of 600 mg (2 tablets of 300 mg) twice daily with food (equivalent to a daily dose of 1200 mg) will be administered orally.
Drug: Goserelin — Goserelin at a dose of 3.6 mg will be administered subcutaneously every 4 weeks.
  Arms: Darolutamide plus Goserelin

SUMMARY:
This study is an open-label phase 2 study to evaluate the safety and efficacy of Darolutamide monotherapy in patients with androgen receptor-positive salivary gland carcinoma. Moreover, this study will evaluate the safety and efficacy of Darolutamide and Goserelin combination in patients with androgen receptor-positive salivary gland carcinoma.

ELIGIBILITY:
Inclusion Criteria:

Darolutamide monotherapy group:

1. Signed, written informed consent.
2. Patients older than 20 years.
3. Histologically confirmed any salivary duct carcinoma (SDC), adenocarcinoma (AC)(NOS), or Carcinoma ex pleomorphic adenoma.
4. Patients with locally recurrent(unresectable) or metastatic salivary gland carcinoma who are not applied for surgery or radiation treatment.
5. Presence of measurable or evaluable disease according to RECIST v1.1
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
7. Adequate organ or bone marrow function
8. Patients who agree to practice effective barrier contraception and refrain from sperm donation during the entire study treatment period and 3 months after the last dose of the study drug.

Darolutamide and Goserelin combination therapy group:

1. Signed, written informed consent.
2. Patients older than 20 years.
3. Histologically confirmed as androgen receptor-positive salivary gland carcinoma at the medical institution.
4. Histologically confirmed as salivary gland carcinoma at the medical institution.
5. Patients with locally recurrent(unresectable) or metastatic salivary gland carcinoma who are not applied for surgery or radiation treatment.
6. Presence of measurable or evaluable disease according to RECIST v1.1
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
8. Adequate organ or bone marrow function
9. Patients who agree to practice effective barrier contraception refrain from sperm donation and stop breastfeeding during the entire study treatment period and through 3 months after the last dose of the study drug.

Exclusion Criteria:

Darolutamide monotherapy group:

1. Histologically confirmed as androgen receptor-negative salivary gland carcinoma at a central laboratory.
2. Prior treatment with AR inhibitors, CYP17 enzyme inhibitors, or LH-RH analogue.
3. Metastases in the brain/central nervous system (CNS).
4. Patients who are pregnant or breastfeeding.
5. Synchronous or metachronous malignancies.
6. Participant has a known history of HIV infection.
7. A positive test result for any of the followings:

   * HBsAg positive
   * HBsAb positive and hepatitis B virus (HBV)-DNA positive
   * HBcAb positive and HBV-DNA positive
8. Severe or uncontrolled concurrent heart disease or hypertension.
9. Inability to swallow oral medications.

Darolutamide and Goserelin combination therapy group:

1. Prior treatment with AR inhibitors, CYP17 enzyme inhibitors, LH-RH analogue, Sex Hormones, or Gonadotropin
2. Prior treatment with Darolutamide or Goserelin.
3. Metastases in the brain/CNS.
4. Patients who are pregnant or breastfeeding.
5. Synchronous or metachronous malignancies.
6. Participant has a known history of HIV infection.
7. A positive test result for any of the followings:

   * HBsAg positive
   * HBsAb positive and HBV-DNA positive
   * HBcAb positive and HBV-DNA positive
8. Severe or uncontrolled concurrent heart disease or hypertension.
9. Inability to administer Darolutamide or Goserelin.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2020-04-17 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Darolutamide monotherapy group: Objective response rate(ORR) assessed by investigators | Up to 13 month
  The proportion of patients with confirmed tumor response of complete response (CR) or partial response (PR) per RECIST 1.1, as assessed by investigators
Darolutamide and Goserelin combination therapy group: Objective response rate(ORR) assessed by an Independent Review Committee | Up to 13 month
  The proportion of patients with confirmed tumor response of CR or PR per RECIST 1.1, as assessed by an independent review committee

SECONDARY OUTCOMES:
Duration of Response (DOR) | Up to 13 month
  DOR will be defined among responders from the date of initial documentation of a response (CR or PR) to the date of first documented evidence of progressive disease as defined in RECIST version 1.1 or death, whichever occurred first.
Best Overall Response (BOR) | Up to 13 month
  BOR will be defined as the best response recorded from the start of protocol treatment based on RECIST version 1.1
Disease Control Rate (DCR) | Up to 13 month
  DCR will be defined as the percentage of participants who achieved a confirmed best overall response of CR, PR, or SD for at least 6 weeks based on RECIST version 1.1.
Clinical Benefit Rate (CBR) | Up to 13 month
  CBR will be defined as the percentage of participants who achieved a confirmed best overall response of CR, PR, or stable disease (SD) for at least 24 weeks based on RECIST version 1.1.
Clinical Benefit Duration (CBD) | Up to 13 month
  CBD will be defined the period starting from the date of enrollment (start of treatment) and ending on the earlier of the date of determination of progression, the date of death from any cause, or the end of the study period.
Progression-Free Survival (PFS) | Up to 13 month
  PFS will be defined as the time from the date of the initial dose of study intervention to the date of first documented disease progression as defined in the RECIST version 1.1, or death due to any cause, whichever occurred first.
Overall Survival (OS) | Up to 13 month
  OS will be defined as the time from the date of the initial dose of study intervention to the date of the participant's death
Adverse events | Up to 30 days after the last dose
  All adverse events, adverse events with undeniable causal relationship to the investigational drug, severe adverse events (SAEs) and SAEs with undeniable causal relationship to the investigational drug will be evaluated based on CTCAE version 5.0
Quality of Life assessed using the EuroQol-5Dimention-5Level (EQ-5D-5L) questionnaire | Up to 30 days after the last dose
  Changes from baseline to each time point in health-related quality of life will be measured using the European Quality of Life Five Dimension Five Level Scale Assessment Questionnaire (EQ-5D-5L). The EQ-5D-5L consists of a description and a health assessment. The health description consists of five dimensions (mobility, self-care, normal activities, pain / discomfort, and anxiety / depression), with each dimension identifying five levels of severity [best (1) - worst (5)]. Health assessment is assessed using a visual analogue scale (VAS)([worse (0) - better (100)].
Darolutamide monotherapy group: ORR assessed by an Independent Review Committee | Up to 13 month
  The proportion of patients with confirmed tumor response of CR or PR per RECIST 1.1, as assessed by an independent review committee
Darolutamide and Goserelin combination therapy group: ORR assessed by investigators | Up to 13 month
  The proportion of patients with confirmed tumor response of complete response (CR) or partial response (PR) per RECIST 1.1, as assessed by investigators
Comparison of androgen receptor (AR) test results in Darolutamide and Goserelin combination therapy group | Baseline
  Comparison of AR test results between each institutional and a central assessment
Positivity of Ki-67 in Darolutamide and Goserelin combination therapy group | Baseline
  The proportion of patients who have high expression of Ki-67 by a central assessment

CONTACTS AND LOCATIONS:
Overall Officials: Makoto Tahara, MD, PhD, Study Director — National Cancer Center Hospital East; Naomi Kiyota, MD, PhD, Study Chair — Kobe University Hospital; Susumu Okano, MD, PhD, Study Chair — National Cancer Center Hospital East
Locations (12):
- Japan (12):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Chiba University Hospital, Chiba, Chiba
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Kyushu Medical Center, Fukuoka, Fukuoka
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kobe University Hospital, Kobe, Hyōgo
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Tohoku University Hospital, Sendai, Miyagi
  - Osaka International Cancer Institute, Osaka, Osaka
  - The Jikei University Hospital, Tokyo, Tokyo
  - Tokyo Medical And Dental University Hospital, Tokyo, Tokyo
  - Tokyo Medical University Hospital, Tokyo, Tokyo

IPD SHARING:
Plan to Share IPD: No